CLINICAL TRIAL: NCT06391320
Title: Obesity Queue Database
Status: Recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-212-B
Record Dates: First submitted 2024-03-31; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: other — Observational studies do not involve intervention

SUMMARY:
To establish an obesity specific disease cohort database and form a special disease cohort, so as to provide guarantee for carrying out high-quality real-world clinical research and clinical research.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years with simple obesity. Simple obesity diagnosis criteria: meet one of the following conditions

  1. BMI≥25 kg/m2
  2. Waist circumference for male/female ≥90/80 cm
  3. Waist-to-hip ratio: 0.9 (male); 0.85 (female)

Exclusion Criteria:

* Patients aged 18-75 years with simple obesity. Simple obesity diagnosis criteria: meet one of the following conditions

  1. BMI≥25 kg/m2
  2. Waist circumference for male/female ≥90/80 cm
  3. Waist-to-hip ratio: 0.9 (male); 0.85 (female)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with obesity, aged 18-75 years, who met the diagnostic criteria for simple obesity and did not participate in any drug clinical trials within 3 months prior to inclusion.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI-PDFF intraperitoneal fat content, fasting and postprandial blood glucose, insulin, C-peptide, glycated hemoglobin, body weight, waist circumference, hip circumference | 5 years
  For a specialized outpatient clinic for obesity, follow-ups should be conducted at 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years. During the trial period and the post-trial observation period, relevant safety indicators must be documented, analyzed statistically, and reported.

SECONDARY OUTCOMES:
Intestinal flora components, glucagon, gastrointestinal hormones GLP-1 and GIP, inflammatory immune indicators, etc | 5 years
  For a specialized outpatient clinic for obesity, follow-ups should be conducted at 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years. During the trial period and the post-trial observation period, relevant safety indicators must be documented, analyzed statistically, and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No